CLINICAL TRIAL: NCT03924388
Title: The Effects of Spinal Cord Stimulation on Autonomic Function in People With Spinal Cord Injury
Brief Title: Spinal Cord Stimulation and Autonomic Response in People With SCI.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: International Collaboration on Repair Discoveries (Other)
Responsible Party: Principal Investigator, Aaron Phillips, Assistant Professor, Physiology & Pharmacology, Cardiac Sciences and Clinical Neurosciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB18- 1592
Record Dates: First submitted 2019-03-21; First posted 2019-04-23 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries; Autonomic Dysreflexia; Orthostatic Hypotension, Dysautonomic
Keywords: Transcutaneous Spinal Cord Stimulation; Epidural Spinal Cord Stimulation; Orthostatic Hypotension; Autonomic Dysreflexia; Spinal Cord Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Shy-Drager Syndrome; Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Project 1 and 2: This multi-site open-label exploratory clinical trial (phase IIb) on examination of the effects of non-invasive transcutaneous spinal cord stimulation will take place at University of Calgary and the University of British Clombia, Canada. In a pseudo-randomized controlled 2×2 between-subject factorial design.
  Project 3: This is a multi-site open-label case study exploring the effects of invasive epidural spinal cord stimulation on small number of individuals with SCI who underwent epidural implantation in Canada or abroad.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short-term transcutaneous spinal cord stimulation (Experimental): In Project 1, we will measure the immediate effects of one-hour mid-thoracic and/or lumbosacral transcutaneous stimulation on autonomic function.
  In mid-thoracic stimulation, the self-adhesive cathode electrode with a diameter of 30 mm will be placed on the skin between the TVII and TVIII spinous processes (approximately corresponding to the T8 spinal segment) at the midline over the vertebral column. For lumbosacral stimulation, the cathode will be placed on the skin between the LI and LII spinous processes (approximately corresponding to the L2/3 to S4/5) at the midline over the vertebral column. Two self-adhesive anode electrodes with a size of 5 × 9 cm will be symmetrically located on the skin over the iliac crests. Before and immediately after the stimulation, the outcomes will be measured in 2 positions, supine and ~ 70° upright (adjusted by tilt-up table).
  Interventions: Device: Trnascutaneous electrical spinal cord stimulation.
- Long-term transcutaneous spinal cord stimulation (Experimental): In Project 2, we will measure the effects of one-month stimulation (five one-hour stimulation sessions per week) of mid-thoracic and lumbosacral transcutaneous spinal cord stimulation on autonomic function.
  The electrode placement and duration of stimulation will be identical to Project 1. The outcomes at each time point will be measured in two positions, supine and ~ 70° upright (adjusted by tilt-up table). The cardiovascular outcomes will be measured before, after the last stimulation session. Bladder and bowel function will be assessed weekly.
  Interventions: Device: Trnascutaneous electrical spinal cord stimulation.
- Project 3 (Experimental): For Project 3, only individuals who have previously been implanted with an epidural stimulator will be invited to participate. They will have only one stimulation session. We will not offer participants to undergo implantation surgery.
  Interventions: Device: Epidural spinal cord stimulation

INTERVENTIONS:
Device: Epidural spinal cord stimulation — The measurements will be obtained in 2 positions of supine and ~ 70° upright adjusted by the tilt-up table.
  Arms: Project 3
Device: Trnascutaneous electrical spinal cord stimulation. — The measurements will be obtained in 2 positions of supine and ~ 70° upright adjusted by the tilt-up table.
  Arms: Long-term transcutaneous spinal cord stimulation; Short-term transcutaneous spinal cord stimulation

SUMMARY:
Despite being studied less than half as frequently, autonomic dysfunction is a greater priority than walking again in spinal cord injury. One autonomic condition after spinal cord injury is orthostatic hypotension, where blood pressure dramatically declines when patients assume the upright posture. Orthostatic hypotension is associated with all-cause mortality and cardiovascular incidents as well as fatigue and cognitive dysfunction, and it almost certainly contributes to an elevated risk of heart disease and stroke in people with spinal cord injury. In addition, autonomic dysfunction leads to bladder, bowel, sexual dysfunctions, which are major contributors to reduced quality and quantity of life. Unfortunately, the available options for treating this condition, are primarily limited to pharmacological options, which are not effective and are associated with various side effects. It has been recently demonstrated that spinal cord stimulation can modulate autonomic circuits and improve autonomic function in people living with spinal cord injury. Neuroanatomically, the thoracolumbar sympathetic pathways are the primary spinal cord segments involved in blood pressure control. Recently, a pilot study has been published demonstrating that transcutaneous spinal cord stimulation of thoracolumbar afferents can improve cardiovascular function. However, some studies have shown that lumbosacral transcutaneous spinal cord stimulation can also elicit positive cardiovascular effects. Therefore, there is no consensus on the optimal strategy in order to deliver transcutaneous spinal cord stimulation to improve the function of the autonomic system, and it may be that lumbosacral (i.e. the stimulation site being used most commonly for restoring leg function is sufficient). Another key knowledge gap in terms of transcutaneous spinal cord stimulation is whether or not the current is directly or indirectly activating these spinal circuits. Last but not least, the effects of epidural spinal cord stimulation on the function of cardiovascular, bladder, bowel and sexual system in spinal cord injury have been investigated in no study yet.

AIMS AND HYPOTHESES:

Aim 1. To examine the effects of short-term (one session) transcutaneous spinal cord stimulation on the frequency and severity of episodes of orthostatic hypotension/autonomic dysfunction, and bladder, bowel, and sexual functions. These effects will be compared at two sites of stimulation.

Hypothesis 1.1: Short-term transcutaneous mid-thoracic cord stimulation will mitigate the severity and frequency of orthostatic hypotension/autonomic dysfunction.

Hypothesis 1.2: Lumbosacral transcutaneous spinal cord stimulation will improve bladder, bowel, and sexual functions.

Aim 2. To examine the effects of long-term (one month) transcutaneous spinal cord stimulation on the severity and frequency of orthostatic hypotension/autonomic dysfunction.

Hypothesis 2.1: Long-term stimulation of the mid-thoracic cord will result in sustained improvements in mitigated severity and frequency of orthostatic hypotension/autonomic dysfunction that is not dependent on active stimulation.

Hypothesis 2.2: Long-term lumbosacral transcutaneous spinal cord stimulation will result in sustained improvements in bowel, bladder, and sexual function that is not dependent on active stimulation.

Aim 3: To examine the effects of short-term (one session) epidural spinal cord stimulation on the severity and frequency of orthostatic hypotension/autonomic dysfunction, and bladder, bowel, and sexual functions.

Hypothesis 3.1: Epidural spinal cord stimulation will mitigate the severity and frequency of orthostatic hypotension/autonomic dysfunction and improve bladder, bowel, and sexual function.

Hypothesis 3.3: There is no significant difference between immediate effects of lumbosacral transcutaneous spinal cord stimulation and epidural spinal cord stimulation on bladder, bowel, and sexual function.

For aim 1, 14 participants with spinal cord injury and no implanted electrodes on the spinal cord will be recruited. Participants will randomly receive one-hour stimulation under each of the two stimulation conditions in a crossover manner: Mid-thoracic and Lumbosacral. For aim 2, 28 individuals with spinal cord injury and no implanted electrode will be pseudo-randomized (1:1) to one of two stimulation sites. Participants will receive one-hour stimulation, five sessions per week for four weeks. Cardiovascular and neurological outcomes will be measured before the first stimulation session and after the last stimulation session. For aim 3, 4 participants with spinal cord injury with implanted electrodes on the spinal cord will be recruited to study the immediate effects of invasive epidural spinal cord stimulation.

All outcomes will be measured in two positions: a) Supine, b) ~ 70° upright tilt-test. Additionally, bowel, bladder, and sexual functions in project 2 will be assessed weekly.

DETAILED DESCRIPTION:
STUDY DESIGN AND DURATION Project 1 and 2: This multi-site open-label exploratory clinical trial (phase IIb) on examination of the effects of non-invasive transcutaneous spinal cord stimulation will take place at the University of Calgary and, UBC, Canada. In a pseudo-randomized controlled 2×2 between-subject factorial design.

Project 3: This is a multi-site open-label case study exploring the effects of invasive epidural spinal cord stimulation on a small number of individuals with spinal cord injury who underwent epidural implantation in Canada or abroad.

Duration of study participation for each participant Eligible participants will be enrolled into the study. Four visits (1 screening session and 3 assessment + stimulation sessions) for project 1 and 21 visits during a month (1 "screening" session, 5 "assessment+ stimulation", and 15 "stimulation only" sessions) for Project 2 will be conducted. Eligible participants who are involved in Project 3 will make two separated visits to our laboratory: one screening session and one "assessment + stimulation" session.

Briefly, the study involves the following:

Project 1, 2, and 3, Visit 1: Screening Phase After providing informed consent, participants will be assigned a unique study number and will be then be assessed for study eligibility. Baseline assessments at this phase include a tilt-up test (to confirm orthostatic hypotension), administration of the Montreal Cognitive Assessment Scale, a take-home bladder and bowel diary (to monitor bladder incontinence and frequency of bowel movements), as well as a take-home Bristol Stool Scale (to monitor constipation). Prior to leaving the site, participants will then be equipped with a 24-hour ambulatory blood pressure monitor in order to establish a baseline parameter of severity and frequency of spontaneous episodes of autonomic dysfunction and orthostatic hypotension.

Project 1, Visits 2- 4 Participants that meet preliminary eligibility requirements will undergo baseline measurements including sympathetic skin responses, cerebral blood flow measurement, cardiovascular monitoring and blood tests (to measure catecholamine level in serum before, during, immediately after tilt up test).

Participants will complete questionnaires, which will establish baseline parameters for self-reported assessments of severity and frequency of autonomic dysfunction, bladder incontinence, and neurogenic bowel Score.

In this randomized crossover study, participants will randomly receive one session of mid-thoracic non-invasive transcutaneous spinal cord stimulation, lumbosacral non-invasive transcutaneous spinal cord stimulation or field block anesthesia. Cardiovascular and neurological outcomes will be measured immediately after stimulation. The stimulation sessions will be separated by at least 72 hours to avoid any interference carry-over effects at each stimulation site. non-invasive transcutaneous spinal cord stimulation is approved under protocols: UBC-Protocol 06 24 14 ca; UCLA, CA - IRB# 14-000158-CR- 00002.

Project 2, Visit 1, Screening Phase After providing the informed consent form for this part of the study (long-term application of Non-invasive Transcutaneous Spinal Cord Stimulation), participants will undergo baseline assessment (explained above) to record severity and frequency of spontaneous episodes of autonomic dysfunction and orthostatic hypotension. participants will be asked to participate in stimulation sessions for four consecutive weeks, with five one-hour sessions of stimulation per week.

Project 2, Visit 2: Baseline measurement and first stimulation session Participants will return 72 hours after the screening phase (explained above). All neurological and cardiovascular outcomes will be measured before applying the first stimulation session. Outcomes will be measured in two positions: a) Supine, b) ~ 70° upright tilt-test, executed in a random order. Participants will then be pseudo-randomized (1:1) to one of the stimulation conditions: 1) Mid-thoracic or 2) Lumbosacral stimulation to receive 60-minute stimulation. Total anticipated time is 3-4 hours including set-up and stimulation.

Project 2, Visits 3 to 20: Stimulation sessions Participants will return to the clinic 24 hours after the first stimulation. All stimulation parameters are identical. Total anticipated time is 2 hours including set-up and one-hour of stimulation. No cardiovascular or neurological outcome will be measured during visits 3 to 20. At the end of 6th, 11th, 16th, and 21st stimulation sessions, neurological bowel Score and the Montreal Cognitive Assessment will be performed. Participants will be sent home with bladder, bowel, and sexual function assessment questionnaires.

All visits will include one tilt-up test with no stimulation, and one with the specific stimulation for that condition, executed in a random order.

Project 2, Visit 21: Last stimulation session and post-intervention outcome measurement In the last visit, participants will receive the last stimulation session, and the cardiovascular and neurological outcome will be measured before and immediately after stimulation. Cardiovascular outcomes measured before and after last stimulation session in two positions: a) Supine and b) ~ 70° upright tilt-test, executed in a random order.

Project 3, Visit 2 For invasive epidural spinal cord stimulation, only individuals who have previously been implanted with an epidural stimulator will be invited to participate. Participants will undergo one "assessment + stimulation" session.The the instructions which are approved under protocols UBC-Protocol 06 24 14 ca; Louisville, KY - IRB Number: 14.0738; Minnesota, MN - IRB Number: 4697-B, USA Veteran's Affairs: IRB Number: 16-4115 will be followed. Outcomes will be measured before and immediately after stimulation. Total anticipated time is 3-4 hours including set-up and all assessments which can be completed in one day.

PROCEDURES AND ASSESSMENTS

Project 1, 2, and 3, Visit 1: Screening Phase

A screening assessment to determine study eligibility will be performed during this visit. After the participant has provided informed consent, he/she will be assigned a unique study number and the following information will be collected:

* Inclusion/Exclusion Criteria
* Medical History
* Demographic information
* Weight and height
* Concomitant Medication and Procedures
* Previous allergies and adverse events to medications

The following procedures will be conducted:

* Self-reported American Spinal Injury Association Impairment Scale
* Autonomic assessment of baseline blood pressure and heart rate and orthostatic instability (i.e., Tilt up test)
* Pregnancy test by a Pregnancy Test Kit (Women of Child Bearing Potential)
* Administration of the Montreal Cognitive Assessment.

The following take home material will be provided:

* Bladder and Bowel Diary (to collect three days of information on incontinence and frequency)
* Bristol Stool Scale (to collect 3 days of information on stool consistency) Project 1, Visits 2 to 4, Project 2, Visits 2 & 21, and Project 3, Visit 2

The following information will be collected:

* Confirmation of Eligibility
* Completed Bladder and Bowel Diary provided at Visit 1
* Completed Bristol Stool Scale provided at Visit 1

The following questionnaires will be administered:

* Self-reported assessments of severity and frequency of autonomic dysfunction
* Adverse Events following electrical stimulation
* Bladder incontinence
* Neurogenic bowel Score
* Female Sexual Distress Scale and Female Sexual Function Index, females only
* International Index of Erectile Function-15, males only

The following procedures will be conducted:

* Blood tests to measure Catecholamine level in serum before, during, immediately after tilt up test.
* 24-hour ambulatory blood pressure monitor
* Sympathetic skin responses Test
* Continuous beat-to-beat measurement of Systolic Blood Pressure, Diastolic Blood Pressure, and Mean Blood Pressure from right finger
* Every minute blood pressure from left Brachial artery Project 2, Visits 6, 11, and 16
* Completed Bladder and Bowel Diary provided at Visit 5, 11, and 15
* Completed Bristol Stool Scale provided at Visit 5, 11, and 15
* Self-reported assessments of severity and frequency of autonomic dysfunction
* Bladder incontinence
* Neurogenic bowel Score
* Female Sexual Distress Scale and Female Sexual Function Index, females only
* International Index of Erectile Function-15, males only
* Adverse Events questionnaire following electrical stimulation For all visits other than the screening phase, participants will be asked to abstain from drugs that directly influence their blood pressure, (e.g., midodrine, fludrocortisone, nifedipine).

Patients will also be asked to arrive having not exercised vigorously for the past 24 hours and to have abstained from caffeine, alcohol, cannabis, and withhold medications for the previous 12 hours and to consume a light breakfast. Upon arrival to the laboratory, participants were asked to empty their bladders to minimize the influence of reflex sympathetic activation on peripheral vascular tone.

Non-invasive Transcutaneous Spinal Cord Stimulation The non-invasive transcutaneous spinal cord stimulation will be performed within the scope of the previously approved ethics by UCLA (45). A stimulator will be utilized for one hour of stimulation. Transcutaneous stimulation will be applied using a self-adhesive cathode electrode with a diameter of 30 mm placed on the skin between the TVII and TVIII spinous processes (approximately corresponding to the T8 spinal segment) at the midline over the vertebral column. For lumbosacral non-invasive transcutaneous spinal cord stimulation, the cathode will be placed on the skin between the LI and LII spinous processes (approximately corresponding to the L2/3 to S4/5) at the midline over the vertebral column. Two self-adhesive anode electrodes with a size of 5 × 9 cm will be symmetrically located on the skin over the iliac crests. Based on previous works it is expect that stimulation will be delivered at 30 Hz as monophasic, 1-ms pulses, to provide afferent input to the region of the spinal cord where sympathetic preganglionic neuron cell bodies are located (24). The current will be increased from 10 mA until blood pressure is normalized. Skin temperature will be monitored in the vicinity of the stimulating electrodes with skin temperature probes.

In invasive epidural spinal cord stimulation, the use of use of stimulator is associated with some risks, including lead migration causing changes in stimulation or reduced functional benefit, lead breakage, over or under stimulation, battery failure, persistent pain at stimulation site, unpleasant sensation or motor disturbance, spinal cord pressure at stimulation site, In non-invasive transcutaneous spinal cord stimulation, again, no adverse event is expected as only parameters and electrodes approved by Health Canada will be utilized in this study. Also, skin temperature for potential irritation will be monitored frequently. Stimulation could elicit autonomic dysfunction, however so far autonomic dysfunction has not been directly observed in the published non-invasive transcutaneous spinal cord stimulation studies. Furthermore, cessation in stimulation immediately reduces blood pressure, and blood pressure closely will be measured during procedures. In case of adverse events, the participant's primary physician would be notified as needed.

Subjects who choose to participate in this trial will be required to give a significant commitment to this study without the guarantee of any benefit. The risks associated with this study are warranted in humans because of the potential direct benefit of the study participants and the spinal cord injury community.

Monitoring during experiment Participants will be continuously monitored for any signs of risks or discomfort. As mentioned, cardiovascular signals such as blood pressure and heart rate will be measured frequently. For non-invasive transcutaneous spinal cord stimulation, skin temperature will be additionally measured. If adverse events occur the testing session will be immediately discontinued. If any complications arise, the experiment will be immediately stopped. In addition, the participant's primary care provider will be notified as necessary if serious adverse events occur.

Data from an autonomic assessment of individuals included in ongoing clinical trials at Foothills Medical Centre (Calgary) and Vancouver General Hospital (Vancouver) with invasive epidural spinal cord stimulation or/and non-invasive transcutaneous spinal cord stimulation after spinal cord injury will be analyzed at Phillips Lab at University of Calgary or within ICORD (UBC). Furthermore, individuals who underwent implantation surgery, either at the above-mentioned study centers or elsewhere, (i.e. as part of a clinical trial or as treatment option), will be assessed and analyzed by Dr. Phillips Lab research team or at ICORD.

Finally, Dr. Phillips lab research team will examine individuals (healthy or following spinal cord injury) using transcutaneous stimulation. No invasive procedure will be carried out. All research protocols for the above-mentioned assessments have been previously approved by the respective research ethics boards at the University of Louisville, UCLA, the University of Minnesota, and UBC: UBC-Protocol 06 24 14 ca; Louisville, KY - IRB Number: 14.0738; Minnesota, MN - IRB Number: 4697-B, USA Veteran's Affairs: IRB Number: 16-4115.

ELIGIBILITY:
Inclusion Criteria:

* Age limit for Project 1 and Project 2 is 18-65 years, and age limit for Project 3 is 22-65 years (Based on FDA approval, participants below 22 are not allowed undergo to implantation surgery).
* The volunteer should have >1-year injury, at least 6 months from any spinal surgery
* Underwent electrode implantation surgery before
* Documented presence of cardiovascular dysfunction including the presence of persistent resting blood pressure and/or symptoms of AD/OH.
* Greater than or equal to antigravity strength in deltoids and biceps bilaterally.
* Participants must have documented 3 days of bladder and bowel history prior to their baseline visit.
* Willing to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
* No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing activities.
* Stable management of spinal cord-related clinical issue (spasticity management).
* Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating.
* Sexually active males with female partners of childbearing potential must agree to effective contraception during th eperiod of the tril nad for at least 28 days after completion of treatment.
* Must provide informed consent.

Exclusion Criteria:

* Presence of severe acute medical issue that in the investigator's judgement would adversely affect the participant's participation in the study.
* Recent treatment with OnabotulinumtoxinA into the detrusor muscle (within 9 months of the baseline visit).
* Ventilator dependent
* Clinically significant depression or ongoing drug abuse
* Use of any medication or treatment that in the opinion of the investigator indicates that it is not the best interest of participant to participate in this study
* Indwelling baclofen pump
* Any implanted metal in the trunk or spinal cord under the sites of application of electrodes (between anode and cathode) for those who are allocated to receive NTSCS.
* Severe anemia (Hgb<8 g/dl) or hypovolemia.
* Participant is a member of the investigational team or his /her immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Episodic Blood Pressure Changes, the unit of measurement is mmHg | In project 1 and 3: before stimulation and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  We will monitor beat-to-beat changes of blood pressure by a Finometer. This outcome will be measured in two different positions: supine and 70 degrees upright position.
Cerebral Blood Flow Changes, the unite of measurement is mililitter/(100 gram tissue minute) | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  We will monitor beat-to-beat changes in blood flow by a Finometer. This outcome will be measured in two different positions: supine and 70 degrees upright position.
Heart Rate Changes, the unit is beat per minute (bpm) | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  We will monitor beat-to-beat changes in heart rate by electrocardiography. This outcome will be measured in two different positions: supine and 70 degrees upright position.
Continues Blood Pressure Changes, the unit of measurement is mmHg | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  We will monitor 24 hours of blood pressure changes by 24-hour Ambulatory Blood Pressure Monitoring.

SECONDARY OUTCOMES:
Sympathetic Skin Responses (SSR) Changes, the unit of measurement is mV | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  The Sympathetic Skin Responses will be elicited by stimulation of median and posterior tibial nerve, and recorded bilaterally and simultaneously from both hands and feet to assess the extent of disruption to spinal autonomic pathways. Ten electrical stimuli (duration 0.2 ms; intensity 8-10 mA) will be applied to the left median nerve and left posterior tibial nerve, in random order and with variable and long-time delays to minimize habituation.
Urodynamic Study Changes | Project 2 only: before the first stimulation session and one week, two weeks, three weeks, and four weeks after the first stimulation session.
  Urodynamic study evaluation typically consists of cystometry with water at 37°C and a filling rate of <30 mL per minute through a 6F double lumen catheter with the participant in the supine position. Abdominal pressure will be measured with a 10F intrarectal balloon catheter. Pelvic floor electromyography will be recorded during cystometry with a bipolar wire electrode in the urethral sphincter. Filling will be stopped when the participants have reported a sensation of fullness, at the moment of urine leakage. The bladder outlet obstruction index (BOOI), will be obtained by formulaic calculations: (BOOI = PdetQmax - 2Qmax). Cystometrogram parameters including first sensation, maximum cystometric capacity (MCC), and the presence of detrusor overactivity with or without incontinence will be annotated. Valsalva leak point pressures will be assessed at a minimum volume of 200 mL. Detrusor compliance was calculated using the formula Compliance= Volume at MCC/Pdet at MCC.
Electromyography (EMG) Changes | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  The Electromyography activity of the skeletal muscles will be also recorded from left and right side to confirm that skeletal muscle contractions are not occurring and therefore the pressure responses are not attributed to the skeletal muscle pump of the venous vasculature. Bipolar surface electrodes will be placed bilaterally on large skeletal muscles such as the vastus lateralis (VL), rectus femoris (RF), and medial hamstrings (MH), tibialis anterior (TA), soleus (SOL), and medial gastrocnemius (MG) muscles. EMG has previously been utilized by our team, as approved by the UBC Clinical Research Ethics Board (H12-02945). Measured EMG potentials range between less than 50 μV and up to 30 mV, depending on the muscle under observation. Typical repetition rate of muscle motor unit firing is about 7-20 Hz, depending on the size of the muscle.
American Spinal Injury Association Impairment Scale (AIS) Changes | In project 1 and 3: before and after one hour spinal cord stimulation. Project 2: before the first stimulation session and after the last stimulation session (one month after the first stimulation session).
  Neurological evaluations of participants with spinal cord injury will be performed using the AIS unless available in the participant chart at the discretion of the investigator. Total duration to do the test is ~ 30 minutes at baseline and ~15 minutes for post-intervention measurements. The level and severity of damage to the motor and sensory pathways will be determined using the standard AIS examination.
Orthostatic Tilt Test Changes | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  Upon arrival to the laboratory, participants will be asked to empty their bladder to minimize the influence of reflex sympathetic activation on peripheral vascular tone (total duration: 25 min). In the supine position, participants will be instrumented with a single- lead ECG. Beat-to-beat systolic (SBP), diastolic (DBP), and mean (MAP) blood pressures will be recorded continuously from the right hand (Finometer; Finapres Medical Systems BV, Arnhem, Netherlands), while discrete blood pressures will be taken every minute from the brachial artery (mmHg). Following instrumentation, baseline recordings will be made during a 10-minute supine rest period. Data acquisition will be performed as detailed above. Participants will then be passively moved to approximately 70° upright stand position by the investigators using the tilt table. This position will be maintained for 15 minutes, during which recordings of heart rate and blood pressure will be continued.
Cerebrovascular Structure Changes | Project 2 only: before the first stimulation session and after the last stimulation session (one month after the first stimulation session).
  For each participant, brachial blood pressure will be measured. The followings will be sampled at 1,000 Hz using an analog-to-digital converter interfaced with data acquisition software on a laptop computer: non-invasive beat-by-beat blood pressure measurement via finger photo plethysmography, electrocardiogram, velocity in the left middle cerebral artery (MCAV) and/or right posterior cerebral artery. These arteries will be insonated using a 2 MHz probe mounted on the temporal bone and a fitted head strap. As described in depth elsewhere, the P1 segment of the posterior cerebral artery and middle cerebral artery (MCA) velocities will be insonated. Arteries will be confirmed using ipsilateral common carotid artery compression, ensuring an increase in posterior cerebral artery velocity and decrease in the middle cerebral artery velocity.
Neurocognitive Changes | Project 2 only: before the first stimulation session and one month after the first stimulation session.
  Participants will remain fitted in the same equipment as used for the cerebrovascular assessment. A visual task will be employed to activate the occipital lobe (while measuring posterior cerebral artery blood flow velocity (cm/sec)). Total duration: 15 minutes.
Autonomic Dysreflexia Health-Related Quality of Life (AD-HR QoL) Questionnaire | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  The AD HR-QoL Questionnaire is derived from the original version of the autonomic dysreflexia sub-section of the Autonomic Dysfunction Following Spinal Cord Injury (ADFSCI) questionnaire which was much more comprehensive in order to assess autonomic dysreflexia frequency and severity on a daily basis and specifically when the bladder is full. The ADFSCI questionnaire was created for use in clinical practice and research to assess blood pressure instability and was designed using the Delphi technique by an expert panel experienced in spinal cord injury treatment. The ADFSCI questionnaire is a 24-item self-reported questionnaire. The questionnaire consists of demographics, medications, frequency/severity of symptoms during autonomic dysreflexia and hypotensive events.
Incontinence Quality of Life (I-QoL) Questionnaire | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  The I-QoL Questionnaire is a self-administered, previously validated and reliable disease-specific questionnaire that measures bladder-related QoL in individuals with neurogenic bladder. The questionnaire is formatted as a 22-items divided into 3 sub-scales: 1) avoidance and limiting behaviour (8 items); 2) psycho-social impact (9 items); and 3) social embarrassment (5 items). Scoring is based on a five-point response scale with values ranging from one (extremely) to five (not at all). Scores are then tallied and transformed into a scale score ranging from 0-100 points with higher scores indicating a greater QoL.
Montreal Cognitive Assessment Scale (MoCA) | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  We will use the MoCA, a standardized cognitive evaluation test. We have utilized this evaluation in our previous studies with spinal cord injury individuals and cognitive deficits related to blood pressure fluctuations. MoCA is a well-accepted general screening tool for individuals with mild cognitive dysfunction. The test assesses eight domains of cognitive functioning, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations and orientation. Total scores below 26 (out of a maximum 30) are considered abnormal and suggest presence of cognitive dysfunctions.
Bristol Stool Scale and Neurogenic Bowel Dysfunction (NBD) Score changes | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  The Bristol Stool Scale is a tool designed to classify faeces into seven categories. The NBD score is a measure of both constipation and fecal incontinence and was developed for and validated in the spinal cord injury population. The NBD score is a 10-item symptom-based score for NBD in individuals with spinal cord injury. The maximum total NBD score is 47 points. The interpretation of the total NBD score is very minor NBD (0-6), minor NBD (7-9), moderate NBD (10-13), and severe NBD (≥14).
Catecholamine Levels in Serum, the unit of this measurement is pmol/L | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  Standard hematology and chemistry laboratory blood tests will be collected by a local laboratory three times in each session: before, during, and immediately after tilt up test. The normal range for epinephrine is 0 to 140 pg/mL (764.3 pmol/L).
Sexual Behaviour Changes | In project 1 and 3: before and after one hour spinal cord stimulation. In project 2: 24 hours before the first stimulation session and after the last stimulation session (session 21, 4 weeks after the first session).
  Sexual behaviour changes will be measured by two questionnaires: one for women and one for men. The Questionnaires are • Female Sexual Distress Scale (FSDS) and Female Sexual Function Index (FSFI), females only and International Index of Erectile Function (IIEF)-15, males only.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheel AW, Krassioukov AV, Inglis JT, Elliott SL. Autonomic dysreflexia during sperm retrieval in spinal cord injury: influence of lesion level and sildenafil citrate. J Appl Physiol (1985). 2005 Jul;99(1):53-8. doi: 10.1152/japplphysiol.00154.2005. Epub 2005 Mar 24. PMID 15790691
- [Background] Solinsky R, Bunnell AE, Linsenmeyer TA, Svircev JN, Engle A, Burns SP. Pharmacodynamics and effectiveness of topical nitroglycerin at lowering blood pressure during autonomic dysreflexia. Spinal Cord. 2017 Oct;55(10):911-914. doi: 10.1038/sc.2017.58. Epub 2017 Jun 6. PMID 28585557
- [Background] Phillips AA, Elliott SL, Zheng MM, Krassioukov AV. Selective alpha adrenergic antagonist reduces severity of transient hypertension during sexual stimulation after spinal cord injury. J Neurotrauma. 2015 Mar 15;32(6):392-6. doi: 10.1089/neu.2014.3590. Epub 2014 Dec 5. PMID 25093677
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Eigenbrodt ML, Rose KM, Couper DJ, Arnett DK, Smith R, Jones D. Orthostatic hypotension as a risk factor for stroke: the atherosclerosis risk in communities (ARIC) study, 1987-1996. Stroke. 2000 Oct;31(10):2307-13. doi: 10.1161/01.str.31.10.2307. PMID 11022055
- [Background] Squair JW, Phillips AA, Harmon M, Krassioukov AV. Emergency management of autonomic dysreflexia with neurologic complications. CMAJ. 2016 Oct 18;188(15):1100-1103. doi: 10.1503/cmaj.151311. Epub 2016 May 24. No abstract available. PMID 27221275
- [Background] Phillips AA, Ainslie PN, Warburton DE, Krassioukov AV. Cerebral Blood Flow Responses to Autonomic Dysreflexia in Humans with Spinal Cord Injury. J Neurotrauma. 2016 Feb 1;33(3):315-8. doi: 10.1089/neu.2015.3871. Epub 2016 Jan 7. PMID 26077616
- [Background] Phillips AA, Warburton DE, Ainslie PN, Krassioukov AV. Regional neurovascular coupling and cognitive performance in those with low blood pressure secondary to high-level spinal cord injury: improved by alpha-1 agonist midodrine hydrochloride. J Cereb Blood Flow Metab. 2014 May;34(5):794-801. doi: 10.1038/jcbfm.2014.3. Epub 2014 Jan 29. PMID 24473484
- [Background] Illman A, Stiller K, Williams M. The prevalence of orthostatic hypotension during physiotherapy treatment in patients with an acute spinal cord injury. Spinal Cord. 2000 Dec;38(12):741-7. doi: 10.1038/sj.sc.3101089. PMID 11175374
- [Background] Freeman R, Abuzinadah AR, Gibbons C, Jones P, Miglis MG, Sinn DI. Orthostatic Hypotension: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Sep 11;72(11):1294-1309. doi: 10.1016/j.jacc.2018.05.079. PMID 30190008
- [Background] Mathias CJ. Orthostatic hypotension and paroxysmal hypertension in humans with high spinal cord injury. Prog Brain Res. 2006;152:231-43. doi: 10.1016/S0079-6123(05)52015-6. PMID 16198704
- [Background] Sclater A, Alagiakrishnan K. Orthostatic hypotension. A primary care primer for assessment and treatment. Geriatrics. 2004 Aug;59(8):22-7. PMID 15332413
- [Background] Bisharat N, Paz E, Klimov A, Friedberg N, Elias M. Cerebral syncope in a patient with spinal cord injury. Pacing Clin Electrophysiol. 2002 Mar;25(3):372-3. doi: 10.1046/j.1460-9592.2002.00372.x. PMID 11990670
- [Background] Currie KD, Krassioukov AV. A walking disaster: a case of incomplete spinal cord injury with symptomatic orthostatic hypotension. Clin Auton Res. 2015 Oct;25(5):335-7. doi: 10.1007/s10286-015-0309-7. Epub 2015 Aug 12. PMID 26264838
- [Background] Claydon VE, Krassioukov AV. Orthostatic hypotension and autonomic pathways after spinal cord injury. J Neurotrauma. 2006 Dec;23(12):1713-25. doi: 10.1089/neu.2006.23.1713. PMID 17184183
- [Background] Sidorov EV, Townson AF, Dvorak MF, Kwon BK, Steeves J, Krassioukov A. Orthostatic hypotension in the first month following acute spinal cord injury. Spinal Cord. 2008 Jan;46(1):65-9. doi: 10.1038/sj.sc.3102064. Epub 2007 Apr 10. PMID 17420772
- [Background] Carlozzi NE, Fyffe D, Morin KG, Byrne R, Tulsky DS, Victorson D, Lai JS, Wecht JM. Impact of blood pressure dysregulation on health-related quality of life in persons with spinal cord injury: development of a conceptual model. Arch Phys Med Rehabil. 2013 Sep;94(9):1721-30. doi: 10.1016/j.apmr.2013.02.024. Epub 2013 Mar 14. PMID 23499779
- [Background] West CR, Krassioukov AV. Autonomic cardiovascular control and sports classification in Paralympic athletes with spinal cord injury. Disabil Rehabil. 2017 Jan;39(2):127-134. doi: 10.3109/09638288.2015.1118161. Epub 2016 Jan 5. PMID 26729004
- [Background] Phillips AA, Squair JW, Krassioukov AV. Paralympic Medicine: The Road to Rio. J Neurotrauma. 2017 Jun 1;34(11):2001-2005. doi: 10.1089/neu.2016.4715. Epub 2017 Jan 24. PMID 27998237
- [Background] Harris P. Self-induced autonomic dysreflexia ('boosting') practised by some tetraplegic athletes to enhance their athletic performance. Paraplegia. 1994 May;32(5):289-91. doi: 10.1038/sc.1994.50. No abstract available. PMID 8058344
- [Background] Gee CM, West CR, Krassioukov AV. Boosting in Elite Athletes with Spinal Cord Injury: A Critical Review of Physiology and Testing Procedures. Sports Med. 2015 Aug;45(8):1133-42. doi: 10.1007/s40279-015-0340-9. PMID 26009300
- [Background] Wecht JM, Rosado-Rivera D, Handrakis JP, Radulovic M, Bauman WA. Effects of midodrine hydrochloride on blood pressure and cerebral blood flow during orthostasis in persons with chronic tetraplegia. Arch Phys Med Rehabil. 2010 Sep;91(9):1429-35. doi: 10.1016/j.apmr.2010.06.017. PMID 20801263
- [Background] Wu JC, Chen YC, Liu L, Chen TJ, Huang WC, Cheng H, Tung-Ping S. Increased risk of stroke after spinal cord injury: a nationwide 4-year follow-up cohort study. Neurology. 2012 Apr 3;78(14):1051-7. doi: 10.1212/WNL.0b013e31824e8eaa. Epub 2012 Feb 29. PMID 22377807
- [Background] Bell EJ, Agarwal SK, Cushman M, Heckbert SR, Lutsey PL, Folsom AR. Orthostatic Hypotension and Risk of Venous Thromboembolism in 2 Cohort Studies. Am J Hypertens. 2016 May;29(5):634-40. doi: 10.1093/ajh/hpv151. Epub 2015 Aug 25. PMID 26306405
- [Background] Agarwal SK, Alonso A, Whelton SP, Soliman EZ, Rose KM, Chamberlain AM, Simpson RJ Jr, Coresh J, Heiss G. Orthostatic change in blood pressure and incidence of atrial fibrillation: results from a bi-ethnic population based study. PLoS One. 2013 Nov 11;8(11):e79030. doi: 10.1371/journal.pone.0079030. eCollection 2013. PMID 24244409
- [Background] Squair JW, DeVeau KM, Harman KA, Poormasjedi-Meibod MS, Hayes B, Liu J, Magnuson DSK, Krassioukov AV, West CR. Spinal Cord Injury Causes Systolic Dysfunction and Cardiomyocyte Atrophy. J Neurotrauma. 2018 Feb 1;35(3):424-434. doi: 10.1089/neu.2017.4984. Epub 2017 Oct 13. PMID 28599602
- [Background] Woodbury MG, Hayes KC, Askes HK. Intermittent catheterization practices following spinal cord injury: a national survey. Can J Urol. 2008 Jun;15(3):4065-71. PMID 18570710
- [Background] Liu N, Fougere R, Zhou MW, Nigro MK, Krassioukov AV. Autonomic dysreflexia severity during urodynamics and cystoscopy in individuals with spinal cord injury. Spinal Cord. 2013 Nov;51(11):863-7. doi: 10.1038/sc.2013.113. Epub 2013 Sep 24. PMID 24060768
- [Background] Teasell RW, Arnold JM, Krassioukov A, Delaney GA. Cardiovascular consequences of loss of supraspinal control of the sympathetic nervous system after spinal cord injury. Arch Phys Med Rehabil. 2000 Apr;81(4):506-16. doi: 10.1053/mr.2000.3848. PMID 10768544
- [Background] Ho CP, Krassioukov AV. Autonomic dysreflexia and myocardial ischemia. Spinal Cord. 2010 Sep;48(9):714-5. doi: 10.1038/sc.2010.2. Epub 2010 Feb 2. PMID 20125109
- [Background] Eltorai I, Kim R, Vulpe M, Kasravi H, Ho W. Fatal cerebral hemorrhage due to autonomic dysreflexia in a tetraplegic patient: case report and review. Paraplegia. 1992 May;30(5):355-60. doi: 10.1038/sc.1992.82. PMID 1598177
- [Background] Wan D, Krassioukov AV. Life-threatening outcomes associated with autonomic dysreflexia: a clinical review. J Spinal Cord Med. 2014 Jan;37(1):2-10. doi: 10.1179/2045772313Y.0000000098. Epub 2013 Nov 26. PMID 24090418
- [Background] Pires PW, Dams Ramos CM, Matin N, Dorrance AM. The effects of hypertension on the cerebral circulation. Am J Physiol Heart Circ Physiol. 2013 Jun 15;304(12):H1598-614. doi: 10.1152/ajpheart.00490.2012. Epub 2013 Apr 12. PMID 23585139
- [Background] Zheng MM, Phillips AA, Elliott SL, Krassioukov AV. Prazosin: a potential new management tool for iatrogenic autonomic dysreflexia in individuals with spinal cord injury? Neural Regen Res. 2015 Apr;10(4):557-8. doi: 10.4103/1673-5374.155422. No abstract available. PMID 26170812
- [Background] Krassioukov A, Warburton DE, Teasell R, Eng JJ; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of autonomic dysreflexia after spinal cord injury. Arch Phys Med Rehabil. 2009 Apr;90(4):682-95. doi: 10.1016/j.apmr.2008.10.017. PMID 19345787
- [Background] Claydon VE, Steeves JD, Krassioukov A. Orthostatic hypotension following spinal cord injury: understanding clinical pathophysiology. Spinal Cord. 2006 Jun;44(6):341-51. doi: 10.1038/sj.sc.3101855. Epub 2005 Nov 22. PMID 16304564
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Hofstoetter US, Freundl B, Binder H, Minassian K. Common neural structures activated by epidural and transcutaneous lumbar spinal cord stimulation: Elicitation of posterior root-muscle reflexes. PLoS One. 2018 Jan 30;13(1):e0192013. doi: 10.1371/journal.pone.0192013. eCollection 2018. PMID 29381748
- [Background] West CR, Phillips AA, Squair JW, Williams AM, Walter M, Lam T, Krassioukov AV. Association of Epidural Stimulation With Cardiovascular Function in an Individual With Spinal Cord Injury. JAMA Neurol. 2018 May 1;75(5):630-632. doi: 10.1001/jamaneurol.2017.5055. PMID 29459943
- [Background] Aslan SC, Legg Ditterline BE, Park MC, Angeli CA, Rejc E, Chen Y, Ovechkin AV, Krassioukov A, Harkema SJ. Epidural Spinal Cord Stimulation of Lumbosacral Networks Modulates Arterial Blood Pressure in Individuals With Spinal Cord Injury-Induced Cardiovascular Deficits. Front Physiol. 2018 May 18;9:565. doi: 10.3389/fphys.2018.00565. eCollection 2018. PMID 29867586
- [Background] Phillips AA, Squair JW, Sayenko DG, Edgerton VR, Gerasimenko Y, Krassioukov AV. An Autonomic Neuroprosthesis: Noninvasive Electrical Spinal Cord Stimulation Restores Autonomic Cardiovascular Function in Individuals with Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):446-451. doi: 10.1089/neu.2017.5082. Epub 2017 Nov 21. PMID 28967294
- [Background] Wecht JM, Bauman WA. Implication of altered autonomic control for orthostatic tolerance in SCI. Auton Neurosci. 2018 Jan;209:51-58. doi: 10.1016/j.autneu.2017.04.004. Epub 2017 May 3. PMID 28499865
- [Background] Biering-Sorensen F, Craggs M, Kennelly M, Schick E, Wyndaele JJ. International lower urinary tract function basic spinal cord injury data set. Spinal Cord. 2008 May;46(5):325-30. doi: 10.1038/sj.sc.3102145. Epub 2007 Nov 27. PMID 18040278
- [Background] Fougere RJ, Currie KD, Nigro MK, Stothers L, Rapoport D, Krassioukov AV. Reduction in Bladder-Related Autonomic Dysreflexia after OnabotulinumtoxinA Treatment in Spinal Cord Injury. J Neurotrauma. 2016 Sep 15;33(18):1651-7. doi: 10.1089/neu.2015.4278. Epub 2016 Apr 13. PMID 26980078
- [Background] Prevention of thromboembolism in spinal cord injury. Consortium for Spinal Cord Medicine. J Spinal Cord Med. 1997 Jul;20(3):259-83. doi: 10.1080/10790268.1997.11719479. No abstract available. PMID 9261774
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Laughlin MH, Schrage WG. Effects of muscle contraction on skeletal muscle blood flow: when is there a muscle pump? Med Sci Sports Exerc. 1999 Jul;31(7):1027-35. doi: 10.1097/00005768-199907000-00016. PMID 10416565
- [Background] Hubli M, Currie KD, West CR, Gee CM, Krassioukov AV. Physical exercise improves arterial stiffness after spinal cord injury. J Spinal Cord Med. 2014 Nov;37(6):782-5. doi: 10.1179/2045772314Y.0000000232. Epub 2014 Jun 29. PMID 24976366
- [Background] Hubli M, Krassioukov AV. Ambulatory blood pressure monitoring in spinal cord injury: clinical practicability. J Neurotrauma. 2014 May 1;31(9):789-97. doi: 10.1089/neu.2013.3148. Epub 2014 Jan 30. PMID 24175653
- [Background] Contributors:; Krassioukov A, Biering-Sorensen CF, Donovan W, Kennelly M, Kirshblum S, Krogh K, Alexander MS, Vogel L, And Wecht J. International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI), First Edition 2012. Top Spinal Cord Inj Rehabil. 2012 Summer;18(3):282-96. doi: 10.1310/sci1803-282. No abstract available. PMID 23460763
- [Background] West CR, Gee CM, Voss C, Hubli M, Currie KD, Schmid J, Krassioukov AV. Cardiovascular control, autonomic function, and elite endurance performance in spinal cord injury. Scand J Med Sci Sports. 2015 Aug;25(4):476-85. doi: 10.1111/sms.12308. Epub 2014 Aug 31. PMID 25175825
- [Background] Costa P, Perrouin-Verbe B, Colvez A, Didier J, Marquis P, Marrel A, Amarenco G, Espirac B, Leriche A. Quality of life in spinal cord injury patients with urinary difficulties. Development and validation of qualiveen. Eur Urol. 2001 Jan;39(1):107-13. doi: 10.1159/000052421. PMID 11173948
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Malhotra A, Shah N, Depasquale J, Baddoura W, Spira R, Rector T. Use of Bristol Stool Form Scale to predict the adequacy of bowel preparation - a prospective study. Colorectal Dis. 2016 Feb;18(2):200-4. doi: 10.1111/codi.13084. PMID 26268220
- [Background] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850